CLINICAL TRIAL: NCT03445208
Title: An Open-Label, Single-Dose, Fixed-Sequence Crossover Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986036 Administered to the Abdomen and Upper Arm in Healthy Participants
Brief Title: A Study of Experimental Medication BMS-986036 Given to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MB130-070
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Hepatic Cirrhosis; Liver Fibrosis; Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease | interventions — Pegbelfermin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): BMI 18.0 to ≤ 25.0
  Interventions: Drug: BMS-986036
- Cohort 2 (Experimental): BMI >25.0 to ≤ 30.0
  Interventions: Drug: BMS-986036
- Cohort 3 (Experimental): BMI >30.0 ≤ 40.0
  Interventions: Drug: BMS-986036

INTERVENTIONS:
Drug: BMS-986036 — Crossover administration to abdomen then upper arm

SUMMARY:
This is a study of experimental medication BMS-986036 given to healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participant, as determined by no clinically significant deviations from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* BMI of 18 to ≤ 40 kg/m2

Exclusion Criteria:

* Presence of any factors that would predispose the participant to infection (eg, extensive periodontal disease that warrants surgical or medical treatment, unhealed open wounds)
* Any bone trauma (fracture) or bone surgery (i.e. hardware placement, joint replacement, bone grafting, or amputation) within 3 months of study drug administration
* Known or suspected autoimmune disorder, excluding vitiligo
* Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status
* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Any major surgery within 6 weeks of study drug administration
* History of diabetes mellitus

Other protocol defined inclusion/exclusion criteria could apply

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) | 29 days
Time of maximum observed serum concentration (Tmax) | 29 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-t)] | 29 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(0-inf)] | 29 days

SECONDARY OUTCOMES:
Number of injection site reactions | Up to 78 days
Number of adverse events (AE) | Up to 78 days
Number of serious adverse events (SAE) | Up to 78 days
Number of AEs leading to discontinuation | Up to 78 days
Number of deaths | Up to 78 days
Serum biomarker antibody concentration | Up to 78 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx